CLINICAL TRIAL: NCT03034733
Title: The Effect of Intravenous Single-dose Dexamethasone on Pain After Total Knee Replacement Surgery
Brief Title: The Effect of Dexamethasone on Pain After Total Knee Replacement Surgery
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Principal investigator (M.K.) left for another workplace. Patient recruitment more difficult than expected.
Sponsor: University of Oulu (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Polvitepdexa 24052016
Record Dates: First submitted 2017-01-03; First posted 2017-01-27 (Estimated); Last update posted 2018-11-29 (Actual); Status verified 2018-11

CONDITIONS: Arthroplasty, Knee Replacement; Pain, Postoperative
Keywords: Arthroplasty; Knee Replacement; Pain, Postoperative; Glucocorticoids; Dexamethasone
MeSH Terms: conditions — Pain, Postoperative | interventions — Dexamethasone; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- dexamethasone 0,15 mg/kg (Experimental): single-dose intravenous dexamethasone 0,15 mg/kg, intraoperative
  Interventions: Drug: Dexamethasone
- dexamethasone 0,25 mg/kg (Experimental): single-dose intravenous dexamethasone 0,25 mg/kg, intraoperative
  Interventions: Drug: Dexamethasone
- Sodium Chloride, (24)NaCl 0,9% (Placebo Comparator): single-dose intravenous saline, intraoperative
  Interventions: Drug: Sodium Chloride, (24)NaCl 0,9%

INTERVENTIONS:
Drug: Dexamethasone — intravenous dexamethasone, two groups: 0,15 mg/kg, 0,25 mg/kg
  Other Names: Oradexon
  Arms: dexamethasone 0,15 mg/kg; dexamethasone 0,25 mg/kg
Drug: Sodium Chloride, (24)NaCl 0,9% — intravenous placebo
  Other Names: saline
  Arms: Sodium Chloride, (24)NaCl 0,9%

SUMMARY:
The purpose of this study is to examine, if a single-dose of dexamethasone given during the operation, alleviates pain after knee replacement surgery.

DETAILED DESCRIPTION:
The purpose of this study is to examine, if a single-dose of dexamethasone given during the operation, alleviates pain after knee replacement surgery. This is also a dose-finding study comparing two doses of dexamethasone.

Total knee arthroplasty causes considerable pain. Multimodal analgesia and peripheral nerve blocks are used for treatment of pain. Some studies suggest that glucocorticoids alleviate postoperative pain. The optimal dose of dexamethasone in treatment of postoperative pain is not known. Studies on this subject in patients with total knee replacement are sparse. Potential side-effects of dexamethasone (hyperglycemia, wound infection) need to be studied.

Patients coming for primary knee replacement surgery are enrolled. The patients in each study group receive multimodal therapy for postoperative pain: etoricoxib, paracetamol, gabapentin and oxycodone. A single dose of intravenous dexamethasone (0,15 mg/kg or 0,25 mg/kg) or a placebo (saline) is administered to the patient during the operation. The effect of dexamethasone on postoperative pain is observed: main outcome is dynamic pain at 24 h postoperatively. The extent of inflammatory reaction is measured (CRP). Serial blood glucose measurements are done.

ELIGIBILITY:
Inclusion Criteria:

* primary total knee replacement surgery
* ASA (american society of anesthesiologists) class 1-3

Exclusion Criteria:

* severe coronary artery disease, heart failure, kidney failure
* insulin-dependent DM (diabetes mellitus), poorly controlled type II DM
* gastric/duodenal ulcer
* allergy/contra-indication for any drug used in the study
* corticosteroid use during last 3 months
* preoperative use of opioid drugs (excl. codeine, tramadol)
* neuropathy/sensory impairment of lower limbs
* lack of co-operation, e.g. inability to use a PCA (patient controlled analgesia)-device

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2017-02-15 (Actual); Primary Completion 2018-01-31 (Actual); Study Completion 2018-01-31 (Actual)

PRIMARY OUTCOMES:
pain during walking, NRS 0-10 | at 24 hours postoperatively
  NRS (numerical rating scale: 0=no pain, 10 = worst possible pain)

SECONDARY OUTCOMES:
pain at rest, NRS 0-10 | preoperatively, postoperatively: at 2 hours, at 8 hours,at 24 hours, at 32 hours, at 48 hours, seventh postoperative day
  NRS (numerical rating scale: 0=no pain, 10 = worst possible pain)
consumption of intravenous oxycodone, milligrams/kilogram body weight | postoperatively: at 2 hours, at 8 hours, at 24 hours, at 48 hours
  cumulative dose of oxycodone administered with a PCA (patient-controlled analgesia)-device
nausea, NRS 0-10 | postoperatively: at 2 hours, at 8 hours,at 24 hours, at 32 hours, at 48 hours
  NRS (numerical rating scale: 0=no nausea, 10 = worst possible nausea)
general wellbeing, NRS 0-10 | postoperatively: at 2 hours, at 8 hours,at 24 hours, at 32 hours, at 48 hours
  NRS (numerical rating scale: 0=worst, 10 = best)
quality of sleep, NRS 0-10 | postoperatively at 24 hours, at 48 hours
  NRS (numerical rating scale: 0=worst, 10 = best)
time to achieve discharge criteria, hours | postoperatively: at 24 hours, at 48 hours, at 72 hours, at 96 hours
  time to achieve discharge criteria, hours
pain during walking, NRS 0-10 | preoperatively, postoperatively: at 8 hours, at 48 hours, seventh postoperative day
  NRS (numerical rating scale: 0=no pain, 10 = worst possible pain)
vomiting, yes/no | postoperatively: at 2 hours, at 8 hours,at 24 hours, at 32 hours, at 48 hours
  vomiting, yes/no

OTHER OUTCOMES:
blood glucose, mmol/l | at preoperative visit, at induction of anesthesia, postoperatively: at 2 hours, at 8 hours, at 24 hours, at 32 hours, at 48 hours
  blood sample
inflammatory reaction, c-reactive protein (CRP) | preoperative, postoperatively: at 24 hours, 48 hours
  blood sample
wound complication, yes/no | postoperatively up to 90 days
  wound complication, yes/no
wound infection, yes/no | postoperatively up to 90 days
  wound infection, yes/no

CONTACTS AND LOCATIONS:
Overall Officials: Matti Kyllönen, MD, Principal Investigator — Oulu University Hospital
Locations (1):
- Oulu University Hospital, Oulu, OYS, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lunn TH, Kehlet H. Perioperative glucocorticoids in hip and knee surgery - benefit vs. harm? A review of randomized clinical trials. Acta Anaesthesiol Scand. 2013 Aug;57(7):823-34. doi: 10.1111/aas.12115. Epub 2013 Apr 15. PMID 23581549
- [Background] Backes JR, Bentley JC, Politi JR, Chambers BT. Dexamethasone reduces length of hospitalization and improves postoperative pain and nausea after total joint arthroplasty: a prospective, randomized controlled trial. J Arthroplasty. 2013 Sep;28(8 Suppl):11-7. doi: 10.1016/j.arth.2013.05.041. Epub 2013 Aug 9. PMID 23937923
- [Background] De Oliveira GS Jr, Almeida MD, Benzon HT, McCarthy RJ. Perioperative single dose systemic dexamethasone for postoperative pain: a meta-analysis of randomized controlled trials. Anesthesiology. 2011 Sep;115(3):575-88. doi: 10.1097/ALN.0b013e31822a24c2. PMID 21799397
- [Background] Gilron I. Corticosteroids in postoperative pain management: future research directions for a multifaceted therapy. Acta Anaesthesiol Scand. 2004 Nov;48(10):1221-2. doi: 10.1111/j.1399-6576.2004.00581.x. No abstract available. PMID 15504179
- [Background] Holte K, Kehlet H. Perioperative single-dose glucocorticoid administration: pathophysiologic effects and clinical implications. J Am Coll Surg. 2002 Nov;195(5):694-712. doi: 10.1016/s1072-7515(02)01491-6. No abstract available. PMID 12437261
- [Background] Husted H, Lunn TH, Troelsen A, Gaarn-Larsen L, Kristensen BB, Kehlet H. Why still in hospital after fast-track hip and knee arthroplasty? Acta Orthop. 2011 Dec;82(6):679-84. doi: 10.3109/17453674.2011.636682. Epub 2011 Nov 9. PMID 22066560
- [Background] Kehlet H. Glucocorticoids for peri-operative analgesia: how far are we from general recommendations? Acta Anaesthesiol Scand. 2007 Oct;51(9):1133-5. doi: 10.1111/j.1399-6576.2007.01459.x. No abstract available. PMID 17850557
- [Background] Koh IJ, Chang CB, Lee JH, Jeon YT, Kim TK. Preemptive low-dose dexamethasone reduces postoperative emesis and pain after TKA: a randomized controlled study. Clin Orthop Relat Res. 2013 Sep;471(9):3010-20. doi: 10.1007/s11999-013-3032-5. Epub 2013 May 4. PMID 23645340
- [Background] Lunn TH, Kristensen BB, Andersen LO, Husted H, Otte KS, Gaarn-Larsen L, Kehlet H. Effect of high-dose preoperative methylprednisolone on pain and recovery after total knee arthroplasty: a randomized, placebo-controlled trial. Br J Anaesth. 2011 Feb;106(2):230-8. doi: 10.1093/bja/aeq333. Epub 2010 Dec 3. PMID 21131371
- [Background] Richards JE, Kauffmann RM, Zuckerman SL, Obremskey WT, May AK. Relationship of hyperglycemia and surgical-site infection in orthopaedic surgery. J Bone Joint Surg Am. 2012 Jul 3;94(13):1181-6. doi: 10.2106/JBJS.K.00193. PMID 22760385
- [Background] Romundstad L, Breivik H, Niemi G, Helle A, Stubhaug A. Methylprednisolone intravenously 1 day after surgery has sustained analgesic and opioid-sparing effects. Acta Anaesthesiol Scand. 2004 Nov;48(10):1223-31. doi: 10.1111/j.1399-6576.2004.00480.x. PMID 15504180
- [Background] Salerno A, Hermann R. Efficacy and safety of steroid use for postoperative pain relief. Update and review of the medical literature. J Bone Joint Surg Am. 2006 Jun;88(6):1361-72. doi: 10.2106/JBJS.D.03018. PMID 16757774
- [Background] Sauerland S, Nagelschmidt M, Mallmann P, Neugebauer EA. Risks and benefits of preoperative high dose methylprednisolone in surgical patients: a systematic review. Drug Saf. 2000 Nov;23(5):449-61. doi: 10.2165/00002018-200023050-00007. PMID 11085349
- [Background] Waldron NH, Jones CA, Gan TJ, Allen TK, Habib AS. Impact of perioperative dexamethasone on postoperative analgesia and side-effects: systematic review and meta-analysis. Br J Anaesth. 2013 Feb;110(2):191-200. doi: 10.1093/bja/aes431. Epub 2012 Dec 5. PMID 23220857
- [Background] Smith C, Erasmus PJ, Myburgh KH. Endocrine and immune effects of dexamethasone in unilateral total knee replacement. J Int Med Res. 2006 Nov-Dec;34(6):603-11. doi: 10.1177/147323000603400605. PMID 17294992
- [Background] Kardash KJ, Sarrazin F, Tessler MJ, Velly AM. Single-dose dexamethasone reduces dynamic pain after total hip arthroplasty. Anesth Analg. 2008 Apr;106(4):1253-7, table of contents. doi: 10.1213/ANE.0b013e318164f319. PMID 18349202